CLINICAL TRIAL: NCT01337960
Title: Ankle Robotics Training After Stroke: Effects on Gait and Balance
Brief Title: Ankle Robotics Training After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: A7461-P
Record Dates: First submitted 2011-04-15; First posted 2011-04-19 (Estimated); Results first posted 2015-06-12 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-05

CONDITIONS: Seated Treadmill Training; Treadmill Locomotor-based Training; Treadmill Only
Keywords: Stroke; Robotics; Neurorehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Experimental): Seated robot training group. Participants at least 6 mos. post-stroke will use the ankle robot in a seated visuo-motor training paradigm. They will train on the robot 3x weekly for 6-weeks (18 sessions) by playing videogames with the paretic ankle. They will be evaluated on outcomes at baseline, post-6 weeks training, and again after a 6-week retention period with no training.
  Interventions: Behavioral: Seated Robot Training (SRT)
- Arm 2 (Experimental): Treadmill training with ankle robot group. Participants at least 6 mos. post-stroke will wear the ankle robot during treadmill locomotor training. They will walk on a treadmill with the ankle robot adjusted to promote paretic ankle engagement during 3 x weekly training sessions over 6 weeks (18 sessions). They will be evaluated on outcomes at baseline, post-6 weeks training, and again after a 6-week retention period with no training.
  Interventions: Behavioral: Treadmill Locomotor-based Training (TMR)
- Arm 3 (Active Comparator): Treadmill only group. This group will consist of participants at least 6 mos. post-stroke who engage in treadmill training 3x weekly for 6 weeks without robotic support. They will be volunteers from another treadmill training study and evaluated on outcomes at baseline and post-6 weeks training. They will not receive retention testing at 12 weeks because they will be continuing with regular treadmill training beyond the 6-week period.
  Interventions: Behavioral: Treadmill Only (TMO)

INTERVENTIONS:
Behavioral: Seated Robot Training (SRT) — Participants at least 6 mos. post-stroke will use the ankle robot in a seated visuo-motor training paradigm. They will train on the robot 3x weekly for 6-weeks (18 sessions) by playing videogames with the paretic ankle. They will be evaluated on outcomes at baseline, post-6 weeks training, and again after a 6-week retention period with no training.
  Arms: Arm 1
Behavioral: Treadmill Locomotor-based Training (TMR) — Treadmill training with ankle robot group. Participants at least 6 mos. post-stroke will wear the ankle robot during treadmill locomotor training. They will walk on a treadmill with the ankle robot adjusted to promote paretic ankle engagement during 3 x weekly training sessions over 6 weeks (18 sessions). They will be evaluated on outcomes at baseline, post-6 weeks training, and again after a 6-week retention period with no training.
  Arms: Arm 2
Behavioral: Treadmill Only (TMO) — Treadmill only group. This group will consist of participants at least 6 mos. post-stroke who engage in treadmill training 3x weekly for 6 weeks without robotic support. They will be volunteers from another treadmill training study and evaluated on outcomes at baseline and post-6 weeks training. They will not receive retention testing at 12 weeks because they will be continuing with regular treadmill training beyond the 6-week period.
  Arms: Arm 3

SUMMARY:
Veterans and other Americans who survive stroke often face disabling motor impairments that impede performance of activities of daily living and limit free-living activity. Prominent among these are diminished walking and balance functions, which not only foster a sedentary lifestyle and physical deconditioning, but also increase the risk of injuries due to falls. Recent research has demonstrated how motor learning based interventions can modify brain activity and improve motor functions in persons with stroke. Now there is a major research opportunity to advance the effectiveness of these interventions by applying new robotics technologies to improve control of essential functions such as gait and balance. One critical area for performance of walking and standing balance is the control of the ankles, as they are a major conduit of mechanical power in gait and also modulate torques affecting the motion of the whole body center of mass when balancing. Thus the current proposal is designed to investigate two approaches for using an impedance controlled ankle robot to improve gait and balance among stroke survivors with chronic lower extremity weakness. One approach uses the ankle robot in a seated visuomotor training program that focuses has subjects play video games with the weaker ankle to improve paretic ankle motor control that may carry over to gait and balance functions. The other approach uses task-specific gait training by integrating use of the ankle robot during treadmill exercise training to assess effects on the same functions. The effectiveness of both robotics approaches will be compared to that of a treadmill exercise program without robotics.

DETAILED DESCRIPTION:
Veterans and other Americans who survive stroke often face disabling motor impairments that impede performance of activities of daily living and limit free-living activity. Prominent among these are diminished locomotor function and impaired balance that not only foster a sedentary lifestyle and physical deconditioning, but also increase the risk injuries due to falls. Recent research has demonstrated how motor learning based interventions can modify brain activity and improve motor functions in persons with stroke. Now there is a major research opportunity to advance the effectiveness of these interventions by applying new robotics technologies to improve neuromotor control of essential functions such as gait and balance. One critical area for performance of walking and standing balance is the control of the ankles, as they are a major conduit of mechanical power in gait and also modulate torques affecting the motion of the whole body center of mass when balancing. Thus the current proposal is designed to investigate two approaches for using an impedance controlled ankle robot to improve gait and balance function among stroke survivors with chronic lower extremity hemiparesis. One approach uses the ankle robot in a seated visuomotor training program that focuses on improving paretic ankle motor control that may transfer to gait and balance functions. The other approach follows the dominant rehabilitation paradigm of task-specific training by integrating use of the ankle robot during treadmill exercise training to assess effects on the same outcomes. The effectiveness of both robotics approaches will be compared to that of a treadmill exercise program without robotics.

The study tests the hypothesis that, in persons with chronic lower extremity hemiparesis, 6 weeks of seated ankle robot training will improve paretic ankle motor control with major improvements in standing balance and moderate improvements in gait, whereas the same amount of training on the treadmill with the ankle robot will improve gait function more than balance. Both robot-trained groups will outperform the treadmill only group on balance, while the treadmill + robot group will make the greatest gains in gait and the seated robot group will make some improvement in gait but will show greater gains in ankle motor control and balance.

Aims: In a 6-week intervention (18 sessions) with persons with chronic lower extremity hemiparesis 1) Compare effects of seated visuomotor ankle robot training vs. treadmill + robot training on paretic ankle impairments and motor control; 2) Compare effects of seated-robot vs. treadmill + robot training on functional mobility and balance outcomes; and 3) Compare the effectiveness of both robotics approaches to a standard treadmill exercise protocol of the same duration. This proposal will establish the initial comparative efficacy of two motor learning based approaches using a modular impedance controlled ankle robot and contrast motor control and functional gait and balance outcomes among them. As a pilot study we also will establish initial deficit profiles for users that respond to each intervention across the 6-week period.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic or hemorrhagic stroke >6 months prior in men or women aged between 18-80 years.
* Clear indications of hemiparetic gait by clinical observation.
* Completed all conventional physical therapy.
* Ability to walk on a treadmill with handrail support.

Exclusion Criteria:

* Cardiac history of (a) unstable angina, (b) recent (less than 3 months) myocardial infarction, congestive heart failure (NYHA category II); (c) hemodynamically significant valvular dysfunction.
* Major clinical depression: CESD score > 16 and judgment of clinical depression
* Medical History: (a) recent hospitalization (less than 3 months) for severe medical disease, (b) symptomatic peripheral arterial occlusive disease, (c) orthopedic or chronic pain conditions that significantly alter gait function, (d) pulmonary or renal failure (e) active cancer
* History of non-stroke neuromuscular disorder restricting gait.
* Aphasia or cognitive functioning that confounds participation, defined as unable to follow 2 step commands. The Mini Mental State Exam will be administered with a cut-off of less than 23 (less than 17 if education level at or below 8th grade), or judgment of the medical officer.
* Hypertension that is a contraindication for a bout of treadmill training (greater than 160/100 on two assessments).
* Self-report of pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-07; Primary Completion 2014-03 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry W Forrester, PhD, Principal Investigator — VA Maryland Health Care System, Baltimore
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Forrester LW, Roy A, Hafer-Macko C, Krebs HI, Macko RF. Task-specific ankle robotics gait training after stroke: a randomized pilot study. J Neuroeng Rehabil. 2016 Jun 2;13(1):51. doi: 10.1186/s12984-016-0158-1. PMID 27255156

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from greater Baltimore area was from IRB approved stroke registry and word of mouth
Pre-assignment Details: Seven subjects who were enrolled (via informed consent) did not receive the allocated intervention due to: relocation (3), lack of transportation (2), re-entry into physical therapy (1), and deemed too high functioning upon neurological re-examination (1). These pre-assignment losses were not counted in the subject tally of baseline assessments.
Groups:
- Seated Robot Training (SRT): Seated robot training group. Participants at least 6 mos. post-stroke will use the ankle robot in a seated visuo-motor training paradigm. They will train on the robot 3x weekly for 6-weeks (18 sessions) by playing videogames with the paretic ankle. They will be evaluated on outcomes at baseline, post-6 weeks training, and again after a 6-week retention period with no training.
  Seated Robot Training (SRT): Participants at least 6 mos. post-stroke will use the ankle robot in a seated visuo-motor training paradigm. They will train on the robot 3x weekly for 6-weeks (18 sessions) by playing videogames with the paretic ankle. They will be evaluated on outcomes at baseline, post-6 weeks training, and again after a 6-week retention period with no training.
- Treadmill Robot Training (TMR): Treadmill training with ankle robot group. Participants at least 6 mos. post-stroke will wear the ankle robot during treadmill locomotor training. They will walk on a treadmill with the ankle robot adjusted to promote paretic ankle engagement during 3 x weekly training sessions over 6 weeks (18 sessions). They will be evaluated on outcomes at baseline, post-6 weeks training, and again after a 6-week retention period with no training.
  Treadmill Locomotor-based Training (TMR): Treadmill training with ankle robot group. Participants at least 6 mos. post-stroke will wear the ankle robot during treadmill locomotor training. They will walk on a treadmill with the ankle robot adjusted to promote paretic ankle engagement during 3 x weekly training sessions over 6 weeks (18 sessions). They will be evaluated on outcomes at baseline, post-6 weeks training, and again after a 6-week retention period with no training.
Period: Overall Study
Arm/Group | Seated Robot Training (SRT) | Treadmill Robot Training (TMR) | Treadmill Only (TMO)
Started | 14 | 14 | 6
Completed | 12 | 14 | 6
Not Completed | 2 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Groups were compared at baseline using Friedmans test and Wilcoxon Sign Rank tests
Groups:
- Total: Total of all reporting groups
Arm/Group | Seated Robot Training (SRT) | Treadmill Robot Training (TMR) | Treadmill Only (TMO) | Total
Number analyzed (Participants) | 14 | 14 | 6 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (13.2) | 59.5 (15.3) | 56.7 (15.2) | 57.8 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 1 | 10
  Male | 10 | 9 | 5 | 24
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 6 | 34

OUTCOME MEASURES:

1. Primary Outcome: Self-selected Floor Walking Velocity Change From Baseline to Post-training and Retention
Description: Velocity and associated spatio-temporal gait parameters from self-selected most comfortable and fastest floor walking over 10m.
Time Frame: Baseline, Post-test training at 6 weeks; Retention at 12 weeks (note TMO control has no retention period)
Population: Nonparametric Fisher's exact test was applied to compare between group changes at retention.
Measure: Mean (Standard Error); unit: cm/sec
Arm/Group | Seated Robot Training (SRT) | Treadmill Robot Training (TMR) | Treadmill Only (TMO)
Number analyzed (Participants) | 12 | 14 | 6
cm/sec
  Baseline | 56.0 (8.3) | 55.5 (5.7) | 50.9 (5.3)
  Post-test Training | 56.1 (8.5) | 58.6 (5.5) | 57.8 (16.5)
  Retention at 12 weeks | 50.9 (7.8) | 61.5 (5.6) | NA (NA) — Controls were in an ongoing treadmill study and could not stop training during the retention period.
Statistical Analysis 1: Comparison: Seated Robot Training (SRT) vs Treadmill Robot Training (TMR); Test type: Superiority or Other; p < 0.01, Fisher Exact

2. Secondary Outcome: Gait Kinetics
Description: Anterior-posterior and medio-lateral ground reaction forces during walking to assess propulsive impulses from paretic and nonparetic sides.
Time Frame: Baseline, Post-test training at 6 weeks; Retention at 12 weeks (note TMO control has no retention period)
Population: Nonparametric Fisher's exact test was applied to compare between group changes at retention.
Measure: Mean (Standard Error); unit: Newton-seconds
Arm/Group | Seated Robot Training (SRT) | Treadmill Robot Training (TMR) | Treadmill Only (TMO)
Number analyzed (Participants) | 12 | 14 | 6
Newton-seconds
  Baseline | 2.1 (4.8) | -2.5 (4.9) | -8.8 (5.9)
  Post-test Training | 0.7 (5.1) | 9.6 (4.1) | -10.1 (6.4)
  Retention at 12 weeks | 4.1 (5.6) | 16.7 (6.0) | NA (NA) — Controls were in an ongoing treadmill study and could not stop training during the retention period.
Statistical Analysis 1: Comparison: Seated Robot Training (SRT) vs Treadmill Robot Training (TMR); Test type: Superiority or Other; p < .02, Fisher Exact

3. Secondary Outcome: Berg Balance Scale
Description: 14-item scale to assess balance function and fall risk, 56 is top score possible (0-56); higher scores indicate higher balance function. Items assess static and dynamic activities of varying difficulty; they are performed to evaluate global level of balance function. Item-level scores range from 0-4, determined by ability to perform the assessed activity; item scores are summed to create the overall score. Subscales are not analyzed.
Time Frame: Baseline, Post-test training at 6 weeks; Retention at 12 weeks (note TMO control has no retention period)
Population: Nonparametric Fisher's exact test was applied to compare between group changes at retention.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Seated Robot Training (SRT) | Treadmill Robot Training (TMR) | Treadmill Only (TMO)
Number analyzed (Participants) | 12 | 14 | 6
units on a scale
  Baseline | 44.3 (3.0) | 49.1 (1.5) | 48.4 (1.9)
  Post-test Training | 45.7 (3.0) | 49.7 (1.5) | 47.4 (2.5)
  12 week Retention | 45.1 (3.6) | 48.8 (1.9) | NA (NA) — Controls were in an ongoing treadmill study and could not stop training during the retention period.
Statistical Analysis 1: Comparison: Seated Robot Training (SRT) vs Treadmill Robot Training (TMR); Test type: Superiority or Other; p = 0.17, Fisher Exact

4. Secondary Outcome: Dynamic Gait Index
Description: The Dynamic Gait Index (DGI) assesses individual's ability to modify balance while walking in the presence of external demands. Performed with a marked distance of 20 feet . The DGI can be performed with or without an assistive device. Scores are based on a 4-point scale: 3 = No gait dysfunction; 2 = Minimal impairment; 1 = Moderate impairment; 0 = Severe impairment. The highest possible score is 24 points. asks include: Steady state walking; Walking with changing speeds; Walking with head turns both horizontally and vertically; Walking while stepping over and around obstacles; Pivoting while walking; Stair climbing.
Time Frame: Baseline, Post-test training at 6 weeks; Retention at 12 weeks (note TMO control has no retention period)
Population: Nonparametric Fisher's exact test was applied to compare between group changes at retention.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Seated Robot Training (SRT) | Treadmill Robot Training (TMR) | Treadmill Only (TMO)
Number analyzed (Participants) | 12 | 14 | 6
units on a scale
  Baseline | 14.4 (1.8) | 17.4 (0.9) | 17.0 (1.1)
  Post-test Training | 16.4 (1.3) | 18.8 (0.8) | 18.4 (1.8)
  Retention at 12 weeks | 17.3 (1.1) | 18.7 (0.9) | NA (NA) — Controls were in an ongoing treadmill study and could not stop training during the retention period.
Statistical Analysis 1: Comparison: Seated Robot Training (SRT) vs Treadmill Robot Training (TMR); Test type: Superiority or Other; p = 0.35, Fisher Exact

5. Secondary Outcome: Anticipatory Postural Adjustments
Description: During gait initiation two force plates measure ground reaction forces and impulses for the postural shifts made in preparation to begin walking.
Time Frame: Baseline, Post-test training at 6 weeks; Retention at 12 weeks (note TMO control has no retention period)
Population: These data were not collected due to technical issues.
Arm/Group | Seated Robot Training (SRT) | Treadmill Robot Training (TMR) | Treadmill Only (TMO)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year, 9 months
Groups:
- Trll Only (TMO): Treadmill only group. This group will consist of participants at least 6 mos. post-stroke who engage in treadmill training 3x weekly for 6 weeks without robotic support. They will be volunteers from another treadmill training study and evaluated on outcomes at baseline and post-6 weeks training. They will not receive retention testing at 12 weeks because they will be continuing with regular treadmill training beyond the 6-week period.
  Treadmill Only (TMO): Treadmill only group. This group will consist of participants at least 6 mos. post-stroke who engage in treadmill training 3x weekly for 6 weeks without robotic support. They will be volunteers from another treadmill training study and evaluated on outcomes at baseline and post-6 weeks training. They will not receive retention testing at 12 weeks because they will be continuing with regular treadmill training beyond the 6-week period.
Arm/Group | Seated Robot Training (SRT) | Treadmill Robot Training (TMR) | Trll Only (TMO)
Serious Adverse Events (participants affected / at risk) | 2/14 | 0/14 | 1/6
Other Adverse Events (participants affected / at risk) | 3/14 | 9/14 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Seated Robot Training (SRT) (N=14) | Treadmill Robot Training (TMR) (N=14) | Trll Only (TMO) (N=6)
Jacksonian Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Subject reported changes in paretic leg function. Immediate screen by study neurologist led to emergency room referral. Subject received complete neuro exam; prescribed antiseizure medication and discharged two days post. Subject completed training.
Ankle sprain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Subject sprained ankle during baseline gait assessment. Returned and completed study.
Chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Subject reported chest pain at home and was seen at local hospital. Report indicated pain was not study related and musculoskeletal in nature.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Seated Robot Training (SRT) (N=14) | Treadmill Robot Training (TMR) (N=14) | Trll Only (TMO) (N=6)
Muscle soreness (Musculoskeletal and connective tissue disorders) | 3 (3) | 7 (13) | 0 (0) — Was more common in early sessions with treadmill + robotics (TMR) as they had more vigorous exercise, resolved in 1-2 days.
Skin abrasion (Skin and subcutaneous tissue disorders) | 0 (0) | 7 (13) | 0 (0) — Early sessions of TMR could evoke excessive rubbing at robot contact points; resolved with extra padding.

LIMITATIONS AND CAVEATS:
The control group was limited in both numbers and the fact that they were not available for retention testing. The technical challenges for reliable collection of anticipatory postural adjustments meant loss of those data for analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes